CLINICAL TRIAL: NCT05237544
Title: Newborn Screening for Spinal Muscular Atrophy (SMA) - a Proof of Principle Study Using Anonymised Blood Spots.
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18NM20
Record Dates: First submitted 2019-06-12; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — All samples used will be leftover dried blood spot material from the Newborn Screening Lab at Great Ormond Street Hospital. . The anonymous known SMA positive blood spots will be provided by an external company (Biogen), in order to determine the accuracy of the assay in detecting SMA positives.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- leftover dried blood spot material: All samples used will be leftover dried blood spot material from the Newborn Screening Lab at Great Ormond Street Hospital.
- anonymous known SMA positive blood spots: The anonymous known SMA positive blood spots will be provided by an external company (Biogen),

SUMMARY:
Spinal muscular atrophy (SMA) is a motor neuron disorder caused by the absence of a functional survival of motor neuron 1, telomeric (SMN1) gene. Type I SMA, a lethal disease of infancy, accounts for the majority of cases. Newborn blood spot screening (NBS)to detect SMA has been implemented in public health laboratories in some countries already. In the UK dried blood spots are collected within a few days of birth on all babies and subsequent newborn screening is currently carried out for other diseases but not for SMA. The investigators would like to carry out a proof of principal testing to show that an assay for SMA can be carried out on these routinely collected dried blood spots (completely anonymised). The investigators would also run some known anonymised SMA positive dried blood spots. The aim is to demonstrate that a simple robust test can be used in a routine diagnostic laboratory to accurately screen for SMA. The investigators will not have access to identifiable data or samples for this project.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a motor neuron disorder caused by the absence of a functional survival of motor neuron 1, telomeric (SMN1) gene. Type I SMA, a lethal disease of infancy, accounts for the majority of cases. The majority of babies born with SMA become symptomatic as babies (type I) or as toddlers (type II). Type I children will never sit unsupported, require ventilated support in the first year of life and usually die before 2 years of age. Type II children can survive to early adulthood but will never walk. They almost invariably develop severe curvature of the spine, feeding and respiratory insufficiency that require appropriate intervention. Cognitive abilities are not impaired and children are generally bright and sociable.

Several new therapies have recently been developed for children with SMA and have shown remarkable success in clinical trials. One of these therapies, spinraza, has received both FDA and EMA approval and is commercially available in most EU countries and in the US, and is being currently evaluated by NICE. Because of the early onset and rapid progression of infantile SMA, prompt detection of the disease is essential to enable successful treatment. It is now recommended that infants be screened for SMA, enabling early drug treatment thus preventing further neuron damage2. The recently published work on the development of spinraza indeed supports the view that children with shorter disease duration had much better outcome [the 2 NEJM papers] a concept that is also emphasised by the interim analysis of infants who received spinraza presymptomatically as part of an ongoing study sponsored by Biogen (Nurture study). The majority of these children had met the age appropriate milestones by the age of 1 year, a clearly remarkable outcome. Similar very promising results were obtained in a recently published AAV gene therapy study in which a number of the severe infants affected by type 1 SMA achieved even the ability to walk unsupported (Mendell SMA gene therapy NEJM 2017). Also in this manuscript, the children who had a shorter disease duration and those treated shortly after the diagnosis had a much better outcome compared to children treated later. While the findings from this early gene therapy study are currently being extended in a larger global phase 3 study, these dramatic results from emerging therapies have led many countries to include SMA in their respective newborn screening programmes.

A previous study (Adams et al. 2014, J. Clin. Imm) was carried out in an almost identical way to the study planned here. The previous study utilised 5000 anonymised leftover blood spots from a routine NBS lab to test the robustness and practicality of running a NBS assay for SCID. This study was scientifically critiqued leading to publication in a respected relevant scientific journal. The study planned here is identical in the approach (5000 normal leftover blood spots) to test the robustness and practicality of using a commercial assay for NBS for SMA in a routine clinical lab environment. As in the previous SCID study we plan to use a number of retrospective known positive samples as well as all the necessary positive/negative controls contained in the commercial kit. The sole aim of the study is to assess the performance of the commercial kit to provide evidence that NBS screening for SMA could feasibly be carried out in routine NBS screening labs.

The investigators therefore believe this is the correct route to take with SMA Newborn Screening as well. Assays for detection of SMA using the dried blood spots collected for Newborn Screening (NBS) have now been developed. This utilises the amplification of the SMN1 gene and subsequent detection of the deleted section that causes SMA. Newborn blood spot screening to detect SMA has been implemented in public health laboratories in some countries already. In the UK, dried blood spots are collected within a few days of birth on all babies and subsequent newborn screening is currently carried out for other diseases but not for SMA.

The investigators would like to carry out a proof of principal testing to show that an assay for SMA can be carried out on these anonymised routinely collected dried blood spots. We would also run some known anonymised SMA positive dried blood spots. The aim is to demonstrate that a simple robust test can be used in a routine diagnostic laboratory to accurately screen for SMA.

ELIGIBILITY:
Inclusion Criteria:

* newborn babies

Exclusion Criteria:

* non-newborn

Ages: 1 Day to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All samples used will be leftover dried blood spot material from the Newborn Screening Lab at Great Ormond Street Hospital. No extra material will be collected and all blood spots will be completely anonymised.
  The anonymous known SMA positive blood spots will be provided by an external company (Biogen), in order to determine the accuracy of the assay in detecting SMA positives.
Sampling Method: Non-Probability Sample
Enrollment: 5065 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of known SMA positive blood spots not detected by NBS | 6 months
  Numbers of false negatives.-This is defined as the number of known SMA positive blood spots not detected by NBS (Newborn Screening).
Ease of use of the assay | 6 months
  Ease of use of the assay in a high-throughput Screening Lab environment. This is defined as the space for equipment and assay set up. It also includes hands-on time setting up and analysing the assay. These are measurable outcomes and will be measured in either dimensions (lab floor/bench space needed) and time (hours) per run.
Number of failed blood spots samples | 6 months
  Number of failed samples. This is defined as the number of blood spots that fail to PCR amplify with the NBS (Newborn Screening) kit.

SECONDARY OUTCOMES:
Assess if the screening assay picks up all known SMA positives | 6 months
  40 SMA positives to be run
Assess if there any false positives with the assay | 6 months
  5000 spots to be run, not expected to be positive

CONTACTS AND LOCATIONS:
Locations (1):
- Dubowitz Neuromuscular Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Adams SP, Gravett E, Kent N, Kricke S, Ifederu A, Scoto M, Samsuddin S, Muntoni F. Screening of Neonatal UK Dried Blood Spots Using a Duplex SMN1 Screening Assay. Int J Neonatal Screen. 2021 Oct 26;7(4):69. doi: 10.3390/ijns7040069. PMID 34842601